CLINICAL TRIAL: NCT06807372
Title: A Multicenter Prospective Study of Artificial Intelligence Predicting Duodenal Stump Leakage After Laparoscopic Radical Gastrectomy for Gastric Cancer
Brief Title: Validation of a Model for Predicting Duodenal Stump Leakage After Gastrectomy
Status: Active, not recruiting | Type: Observational
Sponsor: Jichao Qin (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Jinhua Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Jichao Qin, Professor, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Other Study IDs: 2024-0856
Record Dates: First submitted 2025-02-03; First posted 2025-02-04 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancers
Keywords: artificial intelligence; gastric cancer; duodenal stump leakage; radical gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to validate a machine learning model for predicting duodenal stump leakage after laparoscopic radical gastrectomy for gastric cancer.

DETAILED DESCRIPTION:
Gastrectomy is an essential procedure in radical surgery for gastric cancer. Duodenal stump leakage (DSL) is one of the critical short-term complications after distal and total gastrectomy in gastric cancer patients. Identifying patients with high-risk of DSL will assist the surgeons' decision making to give efficient previous intervention, such as a more rigorous operation, placing dual-lumen flushable drainage catheter and decompression tube in afferent loop. Investigators have developed a high-performance machine learning model based on 4070 gastric cancer patients, which showed good discrimination of DSL. Hence, this multi-center prospective study will validate the reliability of this model for predicting DSL in gastric cancer patients who receive laparoscopic distal or total gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged older than 18 years and younger than 85 years
2. Primary gastric carcinoma confirmed by preoperative pathology result
3. Expected curative resection via laparoscopic distal or total gastrectomy and reconstruction via Billroth-II or Roux-en-Y anastomosis
4. American Society of Anesthesiologists (ASA) class I, II, or III
5. With full documents of preoperative examinations such as blood test and abdominal CT scanning
6. Written informed consent

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Severe mental disorder or language communication disorder.
3. Other surgical procedures of gastrectomy is performed.
4. Interrupted of surgery for more than 30 minutes due to any cause.
5. Malignant tumors with other organs
6. Performed gastrectomy in the past

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves the population of the First Affiliated Hospital of School of Medicine, Zhejiang University, the Second Affiliated Hospital of School of Medicine, Zhejiang University and Jinhua Central Hospital.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of duodenal stump leakage | Within 30 days after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastrointestinal Surgery, The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided